CLINICAL TRIAL: NCT04248621
Title: The Impact of Continuous Versus Intermittent Androgen Deprivation Therapy on Bone Mineral Density Change in Prostate Cancer Patients: A Multicenter, Randomized Clinical Trial
Brief Title: Androgen Deprivation Therapy on Bone Mineral Density Change in Prostate Cancer Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Eulji University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMC 2019-12-003-001
Record Dates: First submitted 2020-01-15; First posted 2020-01-30 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Prostatic Neoplasms
Keywords: Androgen Antagonists; Bone Density; Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Goserelin; Triptorelin Pamoate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; bicalutamide; Flutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Androgen Deprivation (Experimental): ADT including luteinizing hormone-releasing hormone (LHRH) agonist and antagonist, antiandrogen, or maximum androgen blockade (MAB) should be withdrawn after 6 months of ADT, if the prostate-specific antigen (PSA) reaches its nadir (< 4 ng/dL) and serum testosterone reaches castration level (< 50 ng/dL).
  Interventions: Drug: Leuprorelin; Drug: Goserelin; Drug: Triptorelin; Drug: Degarelix; Drug: Bicalutamide; Drug: Flutamide; Drug: Maximum androgen blockade
- Continuous Androgen Deprivation (Active Comparator): ADT including LHRH agonist and antagonist, antiandrogen, or MAB without any discontinuation during study period.
  Interventions: Drug: Leuprorelin; Drug: Goserelin; Drug: Triptorelin; Drug: Degarelix; Drug: Bicalutamide; Drug: Flutamide; Drug: Maximum androgen blockade

INTERVENTIONS:
Drug: Leuprorelin — LHRH agonist
  Other Names: Leuprorelin acetate
Drug: Goserelin — LHRH agonist
  Other Names: Goserelin acetate
Drug: Triptorelin — LHRH agonist
  Other Names: Triptorelin acetate
Drug: Degarelix — LHRH antagonist
  Other Names: Degarelix acetate
Drug: Bicalutamide — Antiandrogen
  Other Names: Casodex
Drug: Flutamide — Antiandrogen
  Other Names: Niftolide
Drug: Maximum androgen blockade — Combination therapy with LHRH agonist and antiandrogen
  Other Names: LHRN agonist and antiandrogen

SUMMARY:
Androgen deprivation therapy (ADT) is a mainstay of prostate cancer treatment to improve overall survival for intermediate- and high-risk localized disease as well as metastatic disease. While ADT improves survival, it can cause significant morbidity and a decrement in quality of life. In particular, ADT is associated with decrease in bone mineral density (BMD) and increased risk of fracture.

Although current guidelines recommend continuous androgen deprivation therapy (CAD) as standard therapy for high-risk disease, there has been increasing recognition of adverse effects from CAD. Since 1986, intermittent androgen deprivation therapy (IAD) as alternative therapeutic strategy for prostate cancer has been proposed to delay development of castration resistance and to reduce the side effects of ADT.

While both CAD and IAD are commonly used in real clinical practice, no prior study examined BMD change after CAD or IAD, and assessed whether bone loss would recover during off-treatment of IAD. The investigators therefore determine the rate of change in BMD induced by ADT (CAD versus IAD) in men with prostate cancer.

DETAILED DESCRIPTION:
Objective: To determine the rate of bone mass loss induced by two therapeutic strategies of ADT (CAD versus IAD) in men with prostate cancer.

Design, setting, and participants: the investigators will perform randomized, open label clinical trial. Men aged over 50 yrs old with prostate cancer (localized, locally advanced, metastatic prostate cancer) who are treated with primary ADT for newly diagnosed prostate cancer or salvage ADT at biochemical recurrence following radical prostatectomy will be included.

Participants will be randomly assigned to one of the following treatment arms:

Arm 1 (CAD): ADT without any discontinuation during study period (12 months).

Arm 2 (IAD): ADT for the first 6 months of study period, if the prostate-specific antigen (PSA) reaches its nadir (< 4 ng/dL) and serum testosterone reaches castration level (< 50 ng/dL).

Outcomes:

Primary outcome: change of L-spine total BMD. Secondary outcomes: change of femur neck BMD, incidence rate of osteoporosis, risk of 10 year major osteoporotic fracture, quality of life based on Expanded Prostate Cancer Index (EPIC) questionnaire.

Timing of outcome measurement: at baseline and up to 12 months after randomization.

Statistical analyses: student's t test for continuous outcomes and Fisher's exact or chi-square test for dichotomous outcomes.

ELIGIBILITY:
Inclusion Criteria:

Men aged over 50 yrs old with histologically diagnosed prostate cancer (localized, locally advanced, metastatic prostate cancer) who are treated with primary ADT for newly diagnosed prostate cancer or salvage ADT at biochemical recurrence following radical prostatectomy. .

Exclusion Criteria:

1. men with double primary malignancies,
2. men who have been treated with ADT or other drug therapy such as denosumab, bisphosphonate or steroid,
3. men with osteoporosis at baseline (T-score ≤ -2.5),
4. men with a known bone disease,
5. men with poor performance status (i.e. Eastern Cooperative Oncology Group performance status 4),
6. men with life expectancy < 12 months,
7. men with increased serum PSA levels (≥ 4 ng/dL) or testosterone levels (≥ 50 ng/dL) even after 6 month ADT,
8. men who are not able to understand trial information or informed consent,

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of L-spine total BMD | At baseline and 12 months
  Measured by bone densitometry

SECONDARY OUTCOMES:
Change of femur neck BMD | At baseline and 12 months
  Measured by bone densitometry
Osteoporosis | At 12 months
  Defined as newly diagnosed osteoporosis based on T-score (≤ -2.5)
Risk of 10 year major osteoporotic fracture | At 12 months
  Estimated by Fracture Risk Assessment Tool (FRAX®, available at www.sheffield.ac.uk/FRAX)
Quality of life after treatment | At baseline and 12 months
  Measured by EPIC questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jinsung Park, MD. PhD., Principal Investigator — Department of Urology, Eulji University, College of Medicine
Locations (10):
- South Korea (10):
  - Department of Urology, Chungbuk National University, College of Medicine, Cheongju-si
  - Department of Urology, Kyungpook National University, School of Medicine, Daegu
  - Department of Urology, Yeungnam University, College of Medicine, Daegu
  - Department of Urology, Eulji University, College of Medicine, Daejeon
  - Department of Urology, Konyang University, College of Medicine,, Daejeon
  - Department of Urology, Chonnam National University, School of Medicine, Gwangju
  - Department of Urology, Wonkwang University, School of Medicine, Iksan
  - Department of Urology,Jeonbuk National University Medical School, Jeonju
  - Department of Urology, Pusan National University, School of Medicine, Pusan
  - Department of Urology, Yonsei University Wonju College of Medicine, Wŏnju

IPD SHARING:
Plan to Share IPD: No